CLINICAL TRIAL: NCT00367796
Title: Genetic Analysis of Craniosynostosis, Philadelphia Type (OMIM 601222)
Brief Title: Genetic Analysis of Craniosynostosis, Philadelphia Type
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999905072; 05-HG-N072
Record Dates: First submitted 2006-08-22; First posted 2006-08-23 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2008-12-23

CONDITIONS: Craniosynostosis; Philadelphia Type Craniosynostosis
Keywords: Craniosynostosis; Philadelphia Type
MeSH Terms: conditions — Craniosynostoses; Craniosynostosis, Philadelphia Type

SUMMARY:
This study will try to find the gene changes responsible for the birth defects in craniosynostosis, Philadelphia type. Craniosynostosis syndromes are a group of conditions that result from closure of one or more of the fibrous joints between the bones of the skull before brain growth is complete. Because of the premature closure, the brain is not able to grow in its natural shape; instead, it compensates with growth in areas of the skull where the joints have not yet closed. The defects in raniosynostosis, Philadelphia type, include skull malformations and webbing of the fingers and toes. Gene changes known to be involved in other craniosynostosis syndromes have not been found in the Philadelphia type syndrome. Therefore, finding the genetic basis of this disorder will provide important new information regarding craniofacial and limb development.

This study includes members of a single large family affected with craniosynostosis, Philadelphia type.

Participants have 1 to 2 teaspoons of blood drawn for genetic studies. A second blood sample may be requested for further research. Some blood may be used to establish a cell line for later studies. This involves growing the white blood cells from the blood sample. The cells can be kept in the laboratory to make more DNA or can be frozen for later use in craniosynostosis studies. Patients may also have their medical records reviewed.

DETAILED DESCRIPTION:
The objective of this study is to determine the molecular basis of craniosynostosis, Philadelphia type. Previous studies by our lab have excluded FGFR1, FGFR2 and FGFR3, the causative genes of most hereditary craniosynostosis syndromes. In the five generation kindred previously reported we have conducted a genome-wide linkage analysis. We have identified four regions linked to this disorder, namely on 2q, 12q, 20q and 22q. Interestingly, syndactyly 1A, a phenotypically similar disorder, demonstrates an overlapping linkage region in two studies. Screening of candidate genes in the redion has excluded ten candidate genes, including IHH, IGFBP2 and IGFBP5.

This protocol is primarily for research purposes. Research subjects may receive benefit from knowing that this research may help other families in the future. Results will be discussed with the primary physician who is a trained medical geneticist. We will emphasize that these are only preliminary findings, that they are not CLIA-approved, and must not be disclosed to the patient or included in the medical record. Repeat testing in a CLIA-approved lab would be required before the specific genetic information could be shared with the patient and family.

ELIGIBILITY:
* INCLUSION CRITERIA:

This research includes only craniosynostosis Philadelphia type patients and members of a single family who were previously referred to us and other family members who have since displayed interest in participating in this study.

EXCLUSION CRITERIA:

Anyone unwilling to provide informed consent (for themselves as adults, or on behalf of their children as minors) or assent.

Medical condition(s) are not in themselves reason for exclusion if in the judgment of the referring physician this would involve no more than minimal risk.

We generally reviewed a brief clinical description from the referring physician about a potential research subject to determine that the subject was appropriate to enter into the study. We reserved the right to exclude cases that were clearly not related to our direct research interests. For new participants, we will review the clinical description from the referring physician and we reserve the right to exclude cases.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2005-01-05; Study Completion 2008-12-23

CONTACTS AND LOCATIONS:
Locations (1):
- Childrens Hospital, Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Robin NH, Segel B, Carpenter G, Muenke M. Craniosynostosis, Philadelphia type: a new autosomal dominant syndrome with sagittal craniosynostosis and syndactyly of the fingers and toes. Am J Med Genet. 1996 Mar 15;62(2):184-91. doi: 10.1002/(SICI)1096-8628(19960315)62:23.0.CO;2-K. PMID 8882401
- [Background] Bosse K, Betz RC, Lee YA, Wienker TF, Reis A, Kleen H, Propping P, Cichon S, Nothen MM. Localization of a gene for syndactyly type 1 to chromosome 2q34-q36. Am J Hum Genet. 2000 Aug;67(2):492-7. doi: 10.1086/303028. Epub 2000 Jun 30. PMID 10877983
- [Background] Ghadami M, Majidzadeh-A K, Haerian BS, Damavandi E, Yamada K, Pasallar P, Najafi MT, Nishimura G, Tomita HA, Yoshiura KI, Niikawa N. Confirmation of genetic homogeneity of syndactyly type 1 in an Iranian family. Am J Med Genet. 2001 Nov 22;104(2):147-51. doi: 10.1002/ajmg.10061. PMID 11746046